CLINICAL TRIAL: NCT03827304
Title: The Development of Interactive Virtual Reality System to Distract Burns Patients Away From Their Pain During Clinical Interventions
Brief Title: Using an Interactive Virtual Reality System to Distract Burns Patients During Burn Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Sheffield (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AA8434
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Burns
Keywords: Burns; Virtual Reality; Qualitative
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: This study aimed to explore:
  * patient and staff perceptions of the effect of active and passive VR on perceived pain and anxiety during painful dressings changes;
  * patient perceptions of the usability, acceptability, engagement with and enjoyment of active and passive VR scenarios;
  * staff perceptions about the usability and implications of the VR technology within a Burns Unit inpatient setting.
  Methods: This was a small-scale qualitative usability study, employing qualitative methods to intervention development and feasibility work.
  Patients: Participants were adult inpatients at the local Burns Unit who were undergoing regular dressing changes during the study period. Exclusion criteria included head and neck burns, wound infection, current diagnosis of PTSD, active psychotic symptoms or high levels of distress. Suitable patients were briefly introduced to the study and supplied with a full information sheet, with details about aims, procedures and rights.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Burns patients (Experimental): This is the group of burns patients that use receive the intervention with the Virtual Reality pain distraction game during the dressing change.
  Interventions: Device: Virtual Reality Distraction for Burns patients

INTERVENTIONS:
Device: Virtual Reality Distraction for Burns patients — Patients wore a VR headset while undergoing a burns dressing change
  Other Names: Burns Dressings Change VR distraction

SUMMARY:
The aims are VR to reduced perceived pain and anxiety during painful dressings changes in a small sample of burns patients;

* to measure the impact of the interventions on objective indicators of pain and distress during dressing changes within the small sample
* to assess pain medication use during virtual reality interventions
* to compare the above effects and experiences across two conditions within each participant: an active version of a virtual reality intervention, and a 'control' condition of no intervention;
* to assess the perceived usability, acceptability, engagement with and enjoyment of the virtual reality intervention to patients
* to consider the apparent feasibility of the virtual reality intervention within a Burns Unit inpatient setting during painful dressing changes 4. Design This is an exploratory feasibility study with a small clinical sample of burns patients and staff caring for them, in a single burns unit setting, employing mixed methods and a repeated measures design to achieve the aims set out above.

DETAILED DESCRIPTION:
The target sample for the clinical feasibility trial are adult burn patients (18+), who were English-speakers, and therefore able to consent for themselves to participate in the research. In order to avoid unnecessary psychological or physical distress, the investigator excluded those with active PTSD or psychotic symptoms, or high levels of distress as judged by Burns Unit clinicians, where the use of VR might be contraindicated. People with mild-moderate or well controlled mental health problems were not be excluded from the study. In addition, those with head and neck burns were excluded as they were unable to wear the VR equipment during dressing changes. The participants were in-patients receiving regular dressing changes during the study period.

Materials used included the VR headset and the software developed using gaming environments, a booklet of questionnaires for the participants to complete, a monitor to measure heart rate, a brief interview schedule, a focus group schedule and digital recording equipment. An active (participatory) gaming environment was developed for participants to trial On three dressing change days participants were asked to complete the two 0-100 ratings 4 times - before their dressing change and three afterwards: immediately after the dressing change and then after 2 and 4 hours. Participants were also asked to complete the scales once on a non-dressing day after the study, to allow assessment of the impact beyond dressing days of the VR intervention. Researcher added in the dates and times for each participant in their booklet. These outcomes were selected as especially important to the study, but also to minimise participant burden. The booklet contained boxes and prompts for participants to add free text responses about the experiences the investigators being monitoring, should participants wish.

Patients were not asked during dressing changes to make any comment about their experience, so that patients could concentrate on the VR environments and to avoid adding to patient burden on the non-intervention condition.

After each VR intervention dressing change, patients were asked a few questions about their experience of pain and the gaming environment, such as 'How was your pain during the dressing change while you were in the VR environment?' 'How did you feel generally during the experience?' 'How helpful did you find the VR during the dressing change?' etc. These short interviews (max 10 minutes) were recorded on a password protected digital recorder.

After both interventions, on a non-dressing change day, another short interview (max 10 minutes) was conducted to enable the participant to make comparisons between the different VR experiences and general comments about their effectiveness, usability and impact compared with no VR. Questions included 'Which VR experience did you prefer and why?' 'From your experience how does a dressing change under VR compare with one with no VR experience?' etc.

Nursing staff were interviewed in a focus group at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* adult burns in-patients
* receiving regular dressing changes during the study period

Exclusion Criteria:

* active PTSD or psychotic symptoms
* high levels of distress
* head and neck burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Phelan, MSc, Principal Investigator — Sheffield Hallam University
Locations (1):
- Ivan Phelan, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will be based on purposive opportunity sampling. People who meet the criteria and are receiving in-patient care during the period of the study.
Groups:
- Burns Dressings Patients: Virtual Reality pain distraction games scenarios
  Virtual Reality Distraction from Burn Pain: Patients wore a VR headset while undergoing a burns dressing change
Period: Overall Study
Arm/Group | Burns Dressings Patients
Started (We aimed to recruit up to 10 participants, in line with similar intervention development and usability studies. However, due to time constraints, we were only able to recruit five patient participants.) | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We aimed to recruit up to 10 participants, in line with similar intervention development and usability studies. However, due to time constraints, we were only able to recruit five patient participants.
Arm/Group | Burns Dressings Patients
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (19.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Using a thermometer scale (Sheffield Burns Unit Psychosocial Screening Tool). Pain was measured on a scale range 0-100 in which 0 is no pain and 100 represents the greatest levels imaginable of pain.
Time Frame: Assessed 1 time during dressing with and without VR
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Burns Patients
Number analyzed (Participants) | 5
score on a scale
  Pain (with VR) | 44.0 (17.1)
  Pain (without VR) | 52.50 (15.54)

2. Secondary Outcome: Anxiety Scores
Description: Using a thermometer scale (Sheffield Burns Unit Psychosocial Screening Tool). Anxiety was measured on a scale range 0-100 in which 0 is no anxiety and 100 represents the greatest levels imaginable of anxiety.
Time Frame: Assessed 1 time during dressing with and without VR
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Burns Dressings Patients
Number analyzed (Participants) | 5
score on a scale
  Anxiety (with VR) | 36.00 (33.61)
  Anxiety (without VR) | 56.25 (31.51)

ADVERSE EVENTS:
Time Frame: A day.
Description: Some people may find the IVR environment disorientating or uncomfortable (e.g. confusion, nausea, dizziness). To avoid any unnecessary discomfort or distress for our participants, we will ensure all those interested in participating have the chance to try out a IVR environment before agreeing to take part. If they feel uncomfortable during the procedure, the IVR can be removed at any stage.
Arm/Group | Burns Dressings Patients
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03827304/Prot_SAP_000.pdf